CLINICAL TRIAL: NCT05654363
Title: The Role of Spinal Analgesia in Laparoscopic and Laparotomic Hysterectomy: an Observational Retrospective Study (the SPIN_GYN Study)
Brief Title: Observational Retrospective Study on Spinal Analgesia in Laparoscopic and Laparotomic Hysterectomy
Acronym: SPIN_GYN
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5421
Record Dates: First submitted 2022-12-05; First posted 2022-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Hysterectomy; Morphine; Anesthesia, Spinal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrathecal morphine: Adult women American Society of Anaesthesiologists (ASA) physical status <= 3, scheduled for elective laparoscopic/laparotomic hysterectomy under general anesthesia between January 1st 2019 and December 31st 2021, who consented to the execution of a preoperative spinal analgesia with intrathecal morphine (as part of our standard practice) and who did not present any contraindications to lumbar puncture.
  Interventions: Procedure: Administration of morphine by intrathecal route
- Intravenous morphine: Adult women American Society of Anaesthesiologists (ASA) physical status <= 3, scheduled for elective laparoscopic/laparotomic hysterectomy under general anesthesia between January 1st 2019 and December 31st 2021, who did not consent to the execution of a preoperative spinal analgesia or presented contraindications to lumbar puncture (coagulopathy or incorrect discontinuation of anticoagulant drugs, increased intracranial pressure, infection at the site of injection, major spinal deformities).
  Interventions: Procedure: Administration of morphine by intravenous route

INTERVENTIONS:
Procedure: Administration of morphine by intrathecal route — Lumbar puncture was performed before the induction of general anesthesia, in the operating room. Spinal anesthesia was performed in sitting position using a midline approach into the L3-L4 or L4-L5 interspaces with a 25ga pencil-point spinal needle administering 75-100 mcg morphine, with or without local anesthetic (levobupivacaine 0,5% 10-15 mg or bupivacaine 0,5% 10-15 mg or ropivacaine 0,5% 10-15 mg), depending on the anesthesiologist's preference. General anesthesia was then conducted according to clinical practice. All patients were transferred in the Post-Anesthesia Care Unit (PACU) at the end of surgery. Throughout the first 48 postoperative hours, all patients were regularly evaluated in the hospital ward by a member of the Acute Pain Service Team.
  Groups: Intrathecal morphine
Procedure: Administration of morphine by intravenous route — General anesthesia was conducted according to clinical practice and a morphine bolus was administered before emergence from anesthesia according to clinical needs. All patients were then transferred in the Post-Anesthesia Care Unit (PACU) at the end of surgery and received Patient-Controlled Analgesia (PCA) with morphine 1mg/mL (CADD®-Solis 2110 Infusion System, Smiths Medical ASD, Inc., USA, 1 mL bolus on demand, no background infusion, 7 minute lockout, max 8 mg/h). Throughout the first 48 postoperative hours, all patients were regularly evaluated in the hospital ward by a member of the Acute Pain Service Team.
  Groups: Intravenous morphine

SUMMARY:
Perioperative multimodal analgesia, defined by the use of various analgesic medications targeting different drug receptors, provides adequate pain relief with minimal or no opiate consumption. Therefore, it represents one of the cornerstone of Enhanced Recovery After Surgery (ERAS) protocols, as the reduction in opioid use and the associated side effects may eventually reduce length of hospital stay, increase patient satisfaction and minimise the risk of long-term opioid use.

Regional and neuraxial anesthesia techniques are key interventions to provide successful analgesia in the context of a multimodal strategy. Intrathecal morphine, for its effectiveness and potential of reducing the need of intravenous postoperative opioids, seems an attractive option in the case of hysterectomy, one of the most common major surgical procedures performed in women, associated with severe postoperative pain even when performed laparoscopically.

The aim of our observational retrospective study is therefore to compare the analgesic efficacy and the safety of morphine administered by intrathecal route versus intravenous route during the first 48 hours after performance of laparoscopic/laparotomic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult women American Society of Anaesthesiologists (ASA) physical status <= 3, scheduled for elective hysterectomy under general anesthesia between January 1st 2019 and December 31st 2021.

Exclusion Criteria:

* patients with American Society of Anaesthesiologists (ASA) status > 3,
* opioid use or history of opioid dependence,
* chronic use of analgesic medications,
* psychiatric disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women American Society of Anaesthesiologists (ASA) physical status <= 3, scheduled for elective hysterectomy under general anesthesia, performed by laparoscopy or by laparotomy (with a Pfannenstiel incision or midline incision).
Sampling Method: Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Time 0 (= baseline, i.e. at the time of Postoperative Anesthesia Care Unit arrival)
  Numeric pain rating scale (NPRS) (ranging from 0, "no pain" and 10, "the worst pain imaginable") at rest
Numeric pain rating scale (NPRS) | 6 hours from baseline
  Numeric pain rating scale (NPRS) (ranging from 0, "no pain" and 10, "the worst pain imaginable") at rest
Numeric pain rating scale (NPRS) | 12 hours from baseline
  Numeric pain rating scale (NPRS) (ranging from 0, "no pain" and 10, "the worst pain imaginable") at rest
Numeric pain rating scale (NPRS) | 24 hours from baseline
  Numeric pain rating scale (NPRS) (ranging from 0, "no pain" and 10, "the worst pain imaginable") at rest
Numeric pain rating scale (NPRS) | 48 hours from baseline
  Numeric pain rating scale (NPRS) (ranging from 0, "no pain" and 10, "the worst pain imaginable") at rest

SECONDARY OUTCOMES:
Adverse events | After the end of surgery, in the first 48 postoperative hours
  Any adverse event, like sedation, itching, nausea, motor weakness, signs of local anesthetic toxicity
Constipation | After the end of surgery, in the first 48 postoperative hours
  The presence of opioid-induced constipation
Mobilization | After the end of surgery, in the first 48 postoperative hours
  Time of first mobilization after the surgical procedure
Intraoperative opioid consumption | During the surgery
  Total opioid consumption
Postoperative opioid consumption | After the end of surgery, in the first 48 postoperative hours
  Total opioid consumption
Rescue analgesia | After the end of surgery, in the first 48 postoperative hours
  The use of non-opioid rescue analgesics in case of NPRS > 3, other than around the clock pain medications
Length of PACU stay | Time from admission to dismissal from PACU, an average of 1 hour
  Length of stay in Postoperative Anesthesia Care Unit (PACU)
Length of hospital stay | Time from dismissal from PACU to dismissal from hospital, an average of 72 hours
  The Length of Hospital Stay (LOS) after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Catarci, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Catarci Stefano, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided